CLINICAL TRIAL: NCT01299896
Title: Connect to Quit: Coordinated Care for Smoking Cessation Among Low Income Veterans
Brief Title: Connect to Quit for Smoking
Acronym: CTQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02936; R01CA141596 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-02-18 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Smoking; Smoking Cessation
Keywords: Cigarette Smoking; Smoking, Tobacco; Tobacco Smoking; Smoking Cessation; Tobacco Dependence
MeSH Terms: conditions — Smoking; Smoking Cessation; Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder | interventions — Smoking Devices; Tobacco Products; Methods; Nicotine Replacement Therapy; Bupropion; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Participants will continue to receive all the care currently offered in the VAPHS, including medications for smoking cessation and use of the in-person or telephone counseling options for quit smoking classes. For veterans with a co-pay, incurred fees with be reimbursed.
  Interventions: Other: Usual Care
- Coordinated Care (Active Comparator): A CTQ Coordinator will coordinate the delivery of smoking related care.
  Interventions: Other: Coordinated Care

INTERVENTIONS:
Other: Coordinated Care — CTQ coordinators will contact the participants for various information sessions about the participant's smoking. These participants will also receive our Connecting to Quit newsletter quarterly.
  Other Names: Smoking, Tobacco; Tobacco Smoking; Smoking Cessation; Tobacco, Intervention; Nicotine Replacement; Buproprion, Wellbutrin; Chantix, Varenicline; Behavorial therapy
  Arms: Coordinated Care
Other: Usual Care — Standard therapy to help participants with smoking cessation.
  Other Names: Smoking, Tobacco; Tobacco Smoking; Smoking Cessation; Tobacco, Intervention; Nicotine Replacement; Buproprion, Wellbutrin; Chantix, Varenicline; Behavorial therapy
  Arms: Usual Care

SUMMARY:
The purpose of this research study is to examine the effectiveness of an intervention designed to reduce smoking in low income veterans within a regional United States Veterans Administration(VA) health care system. A proactive, personalized, coordinated system of care "Connect to Quit (CTQ)" is rooted in the Chronic Care Model. CTQ treats smoking as a chronic condition, like hypertension or diabetes, that requires long term treatment with appropriate combinations of behavioral therapy and pharmacotherapy. CTQ will be evaluated in the context of three (3) VA Pittsburgh Healthcare System (VAPHS) medical practices.

DETAILED DESCRIPTION:
Approximately 40 Primary Care Providers (PCPs), including non-physicians, in the VAPHS and their patients will be recruited and randomized to either Connect to Quit (CTQ) or Usual Care (UC), existing Veterans Health Administration (VHA) services. After PCPs are enrolled, we will begin recruiting their patients who meet eligibility criteria. The desire to quit smoking is not required for participation in the study, as the point of CTQ is to engage smokers at every level of readiness to quit. Target enrollment is 660 participants, approximately 330 in each treatment arm. Participants will be followed for a minimum of 2 years and a maximum of 4. Investigators will measure abstinence (biochemically-validated, 30 day point-prevalence) throughout the study, assessed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Veterans seen by a primary care physician within the VAPHS
* Household income not more than $36,000 annually
* Smoke at least 1 cigarette per day

Exclusion Criteria:

* Smokeless tobacco (snuff or chew) users
* Non-cigarette (e.g., pipe) smokers
* Non-English speaking patients
* Can not be enrolled in another smoking cessation related clinical trial at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary A. Tindle, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Participants will continue to receive all the care currently offered in the Veterans Administration Pittsburgh Healthcare System (VAPHS), including medications for smoking cessation and use of the in-person or telephone counseling options for quit smoking classes. For veterans with a co-pay, incurred fees with be reimbursed.
  Usual Care: Standard therapy to help participants with smoking cessation.
Period: Overall Study
Arm/Group | Usual Care | Coordinated Care
Started | 319 | 314
Completed | 318 | 296
Not Completed | 1 | 18
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Lost to Follow-up | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Coordinated Care | Total
Number analyzed (Participants) | 319 | 314 | 633
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (11.5) | 55.7 (8.7) | 55.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 38 | 66
  Male | 291 | 276 | 567
Region of Enrollment [Number; unit: participants]
  United States | 319 | 314 | 633

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of CTQ vs UC
Description: We will measure abstinence of CTQ smokers vs those in Usual Care (UC). We will biochemically-validate (defined as salivary cotinine <10ng/ml) self reported abstinence (30 day point-prevalence) at the end of 2 years.
Time Frame: Two (2) year period
Measure: Number; unit: percentage of participants per arm
Arm/Group | Usual Care | Coordinated Care
Number analyzed (Participants) | 319 | 314
percentage of participants per arm | 7.5 | 6.1

ADVERSE EVENTS:
Time Frame: Events were collected starting at day 0 and continuing at six month intervals for a minimum of two years maximum 4 years pending date of enrollment.
Description: Hospitalization is the most common serious adverse event for our study population because hospitalization is common among smokers. Serious adverse events were obtained during follow up assessments and/or through chart extraction.
Arm/Group | Usual Care | Coordinated Care
Serious Adverse Events (participants affected / at risk) | 181/319 | 175/314
Other Adverse Events (participants affected / at risk) | 0/319 | 0/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=319) | Coordinated Care (N=314)
Hospitalization (General disorders) | 157 | 162
Death (General disorders) | 24 | 13 (295)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No